CLINICAL TRIAL: NCT01871155
Title: Efficacy Study of Nutri-jelly Intake on Quality of Life in Head and Neck Cancer Patients Undergoing Radiotherapy
Brief Title: Effect of Nutri-jelly on Quality of Life in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dental Innovation Foundation Under Royal Patronage (Other)
Collaborators: Thammasat University (Other); Srinakharinwirot University (Other); Mahidol University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DIF-01
Record Dates: First submitted 2013-05-30; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Cancer; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutri-jelly along with radiotherapy (Experimental): Continuous intake: orally take 1-3 boxes / day for at least 3 days/ week during radiotherapy
  Interventions: Dietary Supplement: Nutri-jelly
- Radiotherapy only (No Intervention): Receive either definitive (total of 30-35 fractions) or palliative ( total of 10 fractions) radiotherapy with no continuous intake of Nutri-Jelly

INTERVENTIONS:
Dietary Supplement: Nutri-jelly — an edible nutritious gel for chewing and swallowing difficulties 1 box contains 250 ml with 250 kcal
  1 serving is considered as food supplement
  Arms: Nutri-jelly along with radiotherapy

SUMMARY:
The purpose of this study is to determine whether a novel edible nutritious gel for patients with chewing and swallowing difficulties, Nutri-jelly, is effective in improving the quality of life of head and neck cancer patients while undergoing conventional radiotherapy.

DETAILED DESCRIPTION:
* independent variable: continuous Nutri -jelly intake
* dependent variable (outcome): changes in health-related quality of life score

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as head and neck cancer
* definitive or palliative radiotherapy treatment plan
* can communicate well

Exclusion Criteria:

* bleeding in the mouth
* respiratory distress
* psychiatric disorders
* radiation field not involve masticatory and swallowing apparatus e.g. certain cases of laryngeal cancer and brain cancer

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes in Health-related quality of life score | 0, 1, 2, 3, 4, 5, 6 weeks after radiotherapy
  * Definitive cases: collect data at baseline (0-5), after Nutri-jelly (6-10), 11-15, 16-20, 21-25, 26-30, 31-35 fractions of RT), total period of 6 weeks
  * Palliative cases: collect data at baseline (0-5), after Nutri-jelly (6-10) fractions of RT, total period of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dunyaporn Trachootham, DDS, PhD, Study Chair — Faculty of Dentistry, Thammasat University, Thailand
Locations (1):
- Mahavachiralongkorn cancer hospital, Pathum Thani, Changwat Pathum Thani, Thailand

REFERENCES:
- See also: Dental Innovation Foundation under royal patronage, His Majesty the King's dental service unit — http://www.dent-in-found.org/